CLINICAL TRIAL: NCT02473471
Title: Micro-osteoperforations and Tooth Movement: A Randomized Controlled Clinical Trial
Brief Title: Micro-osteoperforations and Tooth Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Amal Alkebsi, MClindent in Orthodontics, Department of Preventive Dentistry, Faculty of Dentistry, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JordanUST
Record Dates: First submitted 2015-04-16; First posted 2015-06-16 (Estimated); Results first posted 2017-11-22 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Malocclusion
Keywords: Micro-Osteoperforation (MOPs); regional acceleratory phenomenon (RAP); Malocculsion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MOP side (Experimental): Three small holes in cortical bone can be created by Miniscrews.Before application of the MOPs, Patient will be asked to wash their mouth twice by chlorhexidine for 1 minute. Local anesthesia will be given (2% lidocaine with 1:100,000 epinephrine). Microosteoperforation (MOPs) will be performed distal to canine.
  Interventions: Device: Micro-osteoperforation
- control side (No Intervention): No intervention in the other side of maxilla (control side)

INTERVENTIONS:
Device: Micro-osteoperforation — Three Micro-osteoperforation (MOPs) will be performed distal to canine by Mini screw. Before the application of the MOPs, Patient will be asked to wash their mouth twice by chorhexidine for 1 minute.
  Other Names: Selective alveolar decortication
  Arms: MOP side

SUMMARY:
The purpose of this study is determine the effect the Microosteoperforation (MOPs) using the miniscrew on the rate tooth movement. Moreover, measurement of the level of the pain and pain's interference, the level of satisfaction and comfort using this protocol. Finally root resorption associate with this technique will be evaluated.

DETAILED DESCRIPTION:
This study will be randomized, split mouth design controlled trial with a 1:1 allocation ratio. One resident (A.A), calibrated by the main supervisor (S.M), will be reliable for recruiting the subjects, undertaking the orthodontic treatment under the supervision. The eligibility of the cases will be reevaluated by main supervisor (E.M) before the start of treatment.

Split mouth design will be utilized with MOPs that will be randomly assigned to the patients' left or right sides to eliminate the possibility of uneven occlusal forces because of habitual occlusion predominantly on 1 side and also the eliminate the biological variability between subjects. The allocation sequence will be concealed from the researcher (A.A) enrolling and assessing participants in sequentially numbered, opaque, sealed and stapled envelopes with the participant's the name and date of birth are written before the intervention. Allocation concealment seeks to prevent selection bias, protects the assignment sequence until allocation.

A Ethical approval will be granted by Jordan University of science and technology research center, and permission will be given at postgraduate dental clinics at Jordan University of science and technology, Irbid, Jordan.

We hypothesized that 50% increased in rate of tooth movement in MOP group would produce a clinically significant difference. The sample size was calculated depend on a type I error frequency of 5%. According to the power analysis and assuming a large effect size difference between groups with 50% of acceleration rate of tooth movement, the power analysis yields a total sample size estimate of 44 samples at a conventional alpha-level (p = 0.05) and desired power (1 - β err prob) of 0.90, yielding 22 samples per group (means 22 patients that represent 22 MOP group and 22 Control group). Assuming an overall attrition rate of 15%, initial recruitment should target a total of 55 samples with 18 patients per group. All calculations were performed with the computer application G-Power (Erdfelder et al., 1996)

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* between 16 to 26 years old
* Class II Division 1 malocclusion or bimaxillary protrusion
* Average Lower facial height and Mandibular plane angle
* No systemic disease
* Healthy periodontal condition
* Non smoker
* Probing depth less than 4 mm in all teeth

Exclusion Criteria:

* Long-term use of any Medication
* Poor oral hygiene
* Low and high angle cases
* Systemic disease
* Evidence of bone loss
* Active periodontal disease
* Smoker
* Probing depth more than 4 mm in all teeth

Cephalometric analysis of the included subjects was performed at baseline including

1. Sella-Nasion to A Point Angle (SNA): Measure Description: Sella-Nasion-A point (SNA) indicates the horizontal position of the maxilla relative to the cranial base.
2. Sella-Nasion to B Point Angle (SNB): Sella-Nasion-B point (SNB) indicates the horizontal position of the mandible relative to the cranial base.
3. A point to B Point Angle (ANB): A point- Nasion-B point (ANB) indicates the skeletal relationship between the maxilla and mandible.
4. Maxillary mandibular plane angle (MM): The angle formed between the Maxillary Plane and Mandibular Plane. Maxillary Plane is the plane demonstrated by a line through the anterior and posterior nasal spines.A mandibular plane is a plane demonstrated by a line through the gonion and menton.
5. Lower anterior facial height(LAFH)
6. Upper incisor inclination: The angle between the maxillary plane and the axis of the maxillary incisors.

Ages: 16 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2015-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amal A Alkebsi, MClinDent, Principal Investigator — Jordan University of Science and Technology; Emad Al Maaitah, Ph.D., Principal Investigator — Jordan University of Science and Technology; Hisham Alshorman, Ph.D., Principal Investigator — Jordan University of Science and Technology; Elham S. Abu Alhaija, Ph.D, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Yes
Upon request.
Supporting Information: Study Protocol, SAP
Time Frame: As soon as it published and it to be available anytime.
Access Criteria: Official departments of recognized universities

REFERENCES:
- [Derived] Alkebsi A, Al-Maaitah E, Al-Shorman H, Abu Alhaija E. Three-dimensional assessment of the effect of micro-osteoperforations on the rate of tooth movement during canine retraction in adults with Class II malocclusion: A randomized controlled clinical trial. Am J Orthod Dentofacial Orthop. 2018 Jun;153(6):771-785. doi: 10.1016/j.ajodo.2017.11.026. PMID 29853235

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from a postgraduate clinic at Jordanian University of Science and Technology, in Irbid city, Jordan between Aug 2015 and Jan 2016.
Groups:
- All Study Participants: Split-mouth design study in which the intervention (MOP Side) was randomly assigned to either right or the left side in the maxillary arch where other side serves as a control.
  Randomization was accomplished with block randomization with a permuted block size of 2 with 1:1 allocation ratio to either right or left with allocations concealed in opaque, sealed envelopes. Blinding was applicable at data collection and analysis stage.
Period: Overall Study
Arm/Group | All Study Participants
Started | 35
Received Allocated Intervention | 33
Randomized Not Treated | 2
Completed | 32
Not Completed | 3
Not completed — poor oral hygiene | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Includes groups randomized to receive MOP intervention on one side while the other side serve as control side.
Arm/Group | All Study Participants
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.26 (2.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 10
Region of Enrollment [Number; unit: participants]
  Jordan | 35
Sella-Nasion to A Point Angle (SNA) [Mean (Standard Deviation); unit: Degree] — Sella-Nasion-A point (SNA) indicates the horizontal position of the maxilla relative to the cranial base.
  Degree | 81.9 (4.07)
Sella-Nasion to B Point Angle (SNB) [Mean (Standard Deviation); unit: Degree] — Sella-Nasion-B point (SNB) indicates the horizontal position of the mandible relative to the cranial base.
  Degree | 76.5 (3.85)
A point to B Point Angle (ANB) [Mean (Standard Deviation); unit: Degree] — A point- Nasion-B point (ANB) indicates the skeletal relationship between the maxilla and mandible.
  Degree | 5.5 (2.69)
Maxillary mandibular plane angle [Mean (Standard Deviation); unit: Degree] — The angle formed between the Maxillary Plane and Mandibular Plane.
  Degree | 28.9 (4.27)
Lower anterior facial height(LAFH) [Mean (Standard Deviation); unit: mm] | 55.67 (1.81)
Upper incisor inclination [Mean (Standard Deviation); unit: Degree] — The angle between the maxillary plane and the axis of the maxillary incisors.
  Degree | 119.94 (7.53)

OUTCOME MEASURES:

1. Primary Outcome: 3D Digital Model Measurements of Canine Rate of Tooth Movement
Description: The baseline 3D digital model was superimposed to 3D digital models of the 1st month to determine the anterioposterior displacement of canines.
Time Frame: Baseline to 1st month
Population: Thirty-five subjects were randomized to receive MOP to either right or left sides with 1:1 allocation ratio. Three impressions were missing at first month due to alginate distortion.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- MOP Side: The Micro-osteoperforation side (The Intervention side)
- Control Side: Non intervention side
Arm/Group | MOP Side | Control Side
Number analyzed (Participants) | 29 | 29
mm | 0.65 (0.26) | 0.67 (0.34)
Statistical Analysis 1: Comparison: MOP Side vs Control Side; Test type: Other — The sample size was calculated based on a type I error frequency of 5%. According to the power analysis and assuming a large effect size difference between groups (effect size= 0.8), the power analysis yielded 28 subjects per group at a conventional alpha level (p = 0.05) and desired power (1 - β) of 0.90; p = 0.77, t-test, 2 sided

2. Primary Outcome: 3D Digital Model Measurements of Canine Rate of Tooth Movement
Description: The baseline 3D digital model was superimposed to 3D digital models of 2nd month to determine the anterioposterior displacement of canines.
Time Frame: Baseline to 2nd month
Population: Thirty-five subjects were randomized to receive MOP to either right or left sides with 1:1 allocation ratio. only one impression was lost to be taken by a clinician at two months period.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | MOP Side | Control Side
Number analyzed (Participants) | 31 | 31
mm | 1.36 (0.49) | 1.28 (0.50)
Statistical Analysis 1: Comparison: MOP Side vs Control Side; Test type: Other; p = 0.50, t-test, 2 sided

3. Primary Outcome: 3D Digital Model Measurements of Canine Rate of Tooth Movement
Description: The baseline 3D digital model was superimposed to 3D digital models of 3rd month to determine the anterioposterior displacement of canines.
Time Frame: Baseline to 3rd month
Population: Thirty-five subjects were randomized to receive MOP to either right or left sides with 1:1 allocation ratio. Three impressions were missing at first month due to alginate distortion, and only one impression was lost to be taken by a clinician at two months.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | MOP Side | Control Side
Number analyzed (Participants) | 32 | 32
mm | 1.93 (0.74) | 1.88 (0.67)
Statistical Analysis 1: Comparison: MOP Side vs Control Side; Test type: Other; p = 0.76, t-test, 2 sided

4. Primary Outcome: Intra Oral Measurements of Canine Rate of Tooth Movement
Description: Direct intraoral measurement of the distance between canine and second premolar in the patient's mouth was done every week using a digital caliper, from the upper mesial wing of the canine bracket to upper distal wing of second premolar bracket in both right and left sides parallel to the occlusal plane for 3 months.
Time Frame: Baseline to 1st month
Population: 32 subjects were analyzed to receive MOP to either right or left sides. Only one patient was lost to follow up at the first month time point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | MOP Side | Control Side
Number analyzed (Participants) | 31 | 31
mm | 1.23 (0.45) | 1.17 (0.42)
Statistical Analysis 1: Comparison: MOP Side vs Control Side; Test type: Other; p = 0.56, t-test, 2 sided

5. Primary Outcome: Intra Oral Measurements of Canine Rate of Tooth Movement
Description: as for outcome 4
Time Frame: Baseline to 2nd month
Population: 32 subjects were analyzed to receive MOP to either right or left sides.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | MOP Side | Control Side
Number analyzed (Participants) | 32 | 32
mm | 2.27 (0.72) | 2.24 (0.63)
Statistical Analysis 1: Comparison: MOP Side vs Control Side; Test type: Other; p = 0.88, t-test, 2 sided

6. Primary Outcome: Intra Oral Measurements of Canine Rate of Tooth Movement
Description: as for outcome 4
Time Frame: Baseline to 3 month
Population: 32 subjects were analyzed who received MOP to either right or left sides.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | MOP Side | Control Side
Number analyzed (Participants) | 32 | 32
mm | 3.18 (1.03) | 3.26 (0.81)
Statistical Analysis 1: Comparison: MOP Side vs Control Side; Test type: Other; p = 0.74, t-test, 2 sided — There was no significant difference in tooth movement between control and MOP sides from baseline to 1st, 2nd and 3rd months. P Value < 0.05 was considered statistically significant

7. Secondary Outcome: Root Resorption
Description: It will be evaluated by taking periapical radiograph for canines before canine retraction and after 3 months period
Time Frame: Baseline to 3rd month
Measure: Mean (Standard Deviation); unit: mm
Groups:
- MOP Side: The Micro-osteoperforation side
- Control Side: Non-intervention side
Arm/Group | MOP Side | Control Side
Number analyzed (Participants) | 31 | 31
mm
  Root length at baseline | 19.96 (2.2) | 19.66 (2.5)
  Root length at 3 months | 19.35 (2.0) | 18.93 (2.6)
Statistical Analysis 1: Comparison: MOP Side vs Control Side; Root length at baseline; Test type: Other; p = 0.59, t-test, 2 sided
Statistical Analysis 2: Comparison: MOP Side vs Control Side; Root length at 3 months; Test type: Other; p = 0.48, t-test, 2 sided

8. Secondary Outcome: Pain Intensity
Description: It will be evaluated by using Visual Analog Scale (VAS) from 0 to 10 Numeric Rate Scale in which 0 = no pain and 10 = worst pain.
Time Frame: within 7 days after the intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MOP Side | Control Side
Number analyzed (Participants) | 32 | 32
units on a scale
  Immediate | 1.4 (1.74) | 1.0 (1.99)
  1 hour | 2.4 (2.15) | 1.5 (2.23)
  12 hour | 2.6 (2.79) | 1.6 (2.35)
  Day 1 | 1.2 (1.95) | 0.8 (1.36)
  Day 3 | 0.8 (1.41) | 0.6 (1.29)
  Day 5 | 0.4 (1.10) | 0.3 (1.18)
  Day 7 | 0.2 (0.71) | 0.3 (1.28)
Statistical Analysis 1: Comparison: MOP Side vs Control Side; Immediate after intervention; Test type: Other; p = 0.388, t-test, 2 sided
Statistical Analysis 2: Comparison: MOP Side vs Control Side; 1 hour after intervention; Test type: Other; p = 0.092, t-test, 2 sided
Statistical Analysis 3: Comparison: MOP Side vs Control Side; 12 hour after intervention; Test type: Other; p = 0.100, t-test, 2 sided
Statistical Analysis 4: Comparison: MOP Side vs Control Side; Day 1 after intervention; Test type: Other; p = 0.302, t-test, 2 sided
Statistical Analysis 5: Comparison: MOP Side vs Control Side; Day 3 after intervention; Test type: Other; p = 0.582, t-test, 2 sided
Statistical Analysis 6: Comparison: MOP Side vs Control Side; Day 5 after intervention; Test type: Other; p = 0.743, t-test, 2 sided
Statistical Analysis 7: Comparison: MOP Side vs Control Side; Day 7 after intervention; Test type: Other; p = 0.809, t-test, 2 sided

9. Secondary Outcome: Pain Interference /Pain During Eating?
Description: as for outcome 8
Time Frame: within 7 days after the intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MOP Side | Control Side
Number analyzed (Participants) | 32 | 32
units on a scale
  Day 1 | 3.10 (2.61) | 2.00 (2.54)
  Day 3 | 1.03 (1.58) | 0.65 (1.23)
  Day 5 | 0.29 (0.74) | 0.19 (0.60)
  Day 7 | 0.13 (0.56) | 0.10 (0.54)
Statistical Analysis 1: Comparison: MOP Side vs Control Side; Day 1; Test type: Other; p = 0.09, t-test, 2 sided
Statistical Analysis 2: Comparison: MOP Side vs Control Side; Day 3; Test type: Other; p = 0.29, t-test, 2 sided
Statistical Analysis 3: Comparison: MOP Side vs Control Side; Day 5; Test type: Other; p = 0.57, t-test, 2 sided
Statistical Analysis 4: Comparison: MOP Side vs Control Side; Day 7; Test type: Other; p = 0.82, t-test, 2 sided

10. Secondary Outcome: Pain Interference /Pain Interrupted Sleep
Description: as for outcome 8
Time Frame: within 7 days after the intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MOP Side | Control Side
Number analyzed (Participants) | 31 | 31
units on a scale
  Day 1 | 0.58 (1.69) | 0.19 (0.91)
  Day 3 | 0.13 (0.56) | 0.03 (0.18)
  Day 5 | 0.06 (0.36) | 0.00 (0.00)
  Day 7 | 0.00 (0.00) | 0.00 (0.00)
Statistical Analysis 1: Comparison: MOP Side vs Control Side; Day 1; Test type: Other; p = 0.27, t-test, 2 sided
Statistical Analysis 2: Comparison: MOP Side vs Control Side; Day 3; Test type: Other; p = 0.37, t-test, 2 sided
Statistical Analysis 3: Comparison: MOP Side vs Control Side; Day 5; Test type: Other; p = 0.33, t-test, 2 sided
Statistical Analysis 4: Comparison: MOP Side vs Control Side; Day 7; Test type: Other; p > 0.05, t-test, 2 sided

11. Secondary Outcome: Pain Interference /Swelling of the Surgical Side
Description: It will be evaluated by using Visual Analog Scale (VAS) from 0 to 10 Numeric Rate Scale in which 0 = no swelling and 10 = worst swelling.
Time Frame: within 7 days after the intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MOP Side | Control Side
Number analyzed (Participants) | 31 | 31
units on a scale
  Day 1 | 1.23 (1.68) | 0.41 (1.38)
  Day 3 | 0.48 (1.18) | 0.26 (1.26)
  Day 5 | 0.26 (0.82) | 0.00 (0.00)
  Day 7 | 0.06 (0.25) | 0.00 (0.00)
Statistical Analysis 1: Comparison: MOP Side vs Control Side; Day 1; Test type: Other; p = 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: MOP Side vs Control Side; Day 3; Test type: Other; p = 0.47, t-test, 2 sided
Statistical Analysis 3: Comparison: MOP Side vs Control Side; Day 5; Test type: Other; p = 0.09, t-test, 2 sided
Statistical Analysis 4: Comparison: MOP Side vs Control Side; Test type: Other; p = 0.16, t-test, 2 sided

12. Secondary Outcome: Pain Interference /Discomfort
Description: It will be evaluated by using Visual Analog Scale (VAS) from 0 to 10 Numeric Rate Scale in which 0 = no discomfort and 10 = worst discomfort.
Time Frame: within 7 days after the intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MOP Side | Control Side
Number analyzed (Participants) | 31 | 31
units on a scale
  Day 1 | 2.10 (2.52) | 1.29 (2.19)
  Day 3 | 0.77 (1.36) | 0.58 (1.29)
  Day 5 | 0.23 (0.56) | 0.10 (0.40)
  Day 7 | 0.06 (0.25) | 0.03 (0.18)
Statistical Analysis 1: Comparison: MOP Side vs Control Side; Day 1; Test type: Other; p = 0.18, t-test, 2 sided
Statistical Analysis 2: Comparison: MOP Side vs Control Side; Day 3; Test type: Other; p = 0.57, t-test, 2 sided
Statistical Analysis 3: Comparison: MOP Side vs Control Side; Day 5; Test type: Other; p = 0.30, t-test, 2 sided
Statistical Analysis 4: Comparison: MOP Side vs Control Side; Day 7; Test type: Other; p = 0.56, t-test, 2 sided

13. Secondary Outcome: Patient Satisfaction
Description: It will be evaluated by using Visual Analog Scale (VAS) from 0 to 10 Numeric Rate Scale in which 0 = unsatisfied and 10 = most satisfaction.
Time Frame: After 7 days of MOP application
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MOP Side
Number analyzed (Participants) | 32
units on a scale | 8.94 (1.35)
Statistical Analysis 1: Comparison: MOP Side; Test type: Other; p < 0.05, Descriptive statistics

14. Secondary Outcome: Menstrual Cycle
Description: the relationship between the rate of tooth movement and Menstrual cycle
Time Frame: within 3 months
Population: Sufficient data were not collected from any participant
Arm/Group | MOP Side | Control Side
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months after intervention
Arm/Group | MOP Side | Control Side
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

LIMITATIONS AND CAVEATS:
1. Effect of intervention on inflammatory markers was not evaluated.
2. Short-term clinical study with only 3-months follow up period.
3. Most of the study subjects were females (75%).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-21): https://cdn.clinicaltrials.gov/large-docs/71/NCT02473471/Prot_SAP_000.pdf